CLINICAL TRIAL: NCT06318975
Title: The Effectiveness of Text-Based Messaging Strategies for Preventing Subsequent Problematic Alcohol Use Among Technical Trainees in the US Air Force
Brief Title: Text-Based Messaging Strategies for Preventing Subsequent Problematic Alcohol Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Memphis (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kara Wiseman, MPH, PhD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAPTOR; R01AA029074 (NIH)
Record Dates: First submitted 2024-02-28; First posted 2024-03-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Drinking; Binge Drinking; Text Messaging
Keywords: Military Population Health; Brief Alcohol Intervention; BAI
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Alcohol Intervention (Placebo Comparator): Those assigned to the BAI condition receive the standard BAI, which we have conducted since 2010, during the 4th week of Technical Training, the last week of enforced abstinence. This BAI has become the de-facto standard of care and is part of USAF Training. The BAI is a group-based, one-hour session which includes the following components: Interactive discussion of the positives and negatives of drinking during training and heavy vs. moderate drinking; Discussion of USAF rules on alcohol use and penalties for violations; Discussion of impact of alcohol on military readiness; effects of alcohol and hangover on performance; Review of standard drinks, blood alcohol levels and tolerance; and normative feedback on the Airmen's drinking level compared to others. We will engage in a conversation about whether they have observed concerning patterns of alcohol misuse among other USAF personnel, and how to handle this, along with harm reduction and alcohol refusal strategies.
  Interventions: Behavioral: Brief Alcohol Intervention
- BAI + Texting (Experimental): Those assigned to this arm will receive the same BAI as the other arm with the addition of automated text messages.
  Interventions: Behavioral: Brief Alcohol Intervention; Behavioral: Automated and Targeted Text Messages

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention — All Airmen will receive a standard BAI during the 4th week of Technical Training, the last week of enforced abstinence. The BAI is a group-based, one-hour session which includes the following components: Interactive discussion of the positives and negatives of drinking during training and heavy vs. moderate drinking; Discussion of USAF rules on alcohol use and penalties for violations; Discussion of impact of alcohol on military readiness; effects of alcohol and hangover on performance; Review of standard drinks, blood alcohol levels and tolerance; and normative feedback on the Airmen's drinking level compared to others. We will engage in a conversation about whether they have observed concerning patterns of alcohol misuse among other USAF personnel, and how to handle this, along with harm reduction and alcohol refusal strategies.
Behavioral: Automated and Targeted Text Messages — All messages are pre-written, and their timing is pre-planned - All Airmen will start receiving 3-5 text messages per week starting the Monday after they received the Brief Alcohol Intervention and lasting for six weeks. The intervention is also targeted to age, with some messaging differing for Airmen less than 21 years and those already 21 years old or who will turn 21 during the intervention period. All Airmen randomized to the text message arm will be enroll into the supplemental program, and may opt out at any time. Messages reinforce content of the BAI and provide additional, actionable advice on reducing or avoiding alcohol in more detail and specificity than time typically allows for during the BAI. Messages are sent on days and at times that were indicated as being preferred during formative development of the intervention. Messages are designed to maintain or enhance skill building. No drinking behavior is collected as part of the text messaging intervention
  Arms: BAI + Texting

SUMMARY:
Binge drinking, and its health/social consequences are substantial public health concerns, with a high prevalence in young adults, especially in the US military. Alcohol consumption in the military is very high and normative, but there is zero tolerance for alcohol-related legal trouble, and Air Force Airmen who experience this (e.g., DUI, sexual assault) typically receive a disciplinary action referred to as an Alcohol Related Incident (ARI).

Brief Alcohol Interventions (BAIs) for alcohol misuse are effective in young adults who report binge drinking. Many BAI studies targeted young adults who drink hazardously; these individuals are typically not interested in abstaining but may try decreasing the amount or change the manner in which they drink in order to reduce harmful consequences. The investigators previously published the results of a BAI group-based intervention that reduced ARIs in over 150,000 Airmen on average by 16%. Since 2010, the BAI has been disseminated to most USAF Airmen in Technical Training. However, it is clear additional research is needed to enhance the efficacy of the intervention and reduce risks associated with problem drinking. One strategy to improve health outcomes is well-timed, tailored, and automated text messages. Building on the researchers' preliminary study where text messages reduced driving after drinking as well as total drinks consumed before driving, text messaging may be highly effective when sent at the precise time that Airmen gain access to alcohol (the first time they are allowed off base), a standard time for all Technical Trainees.

One challenge to conducting alcohol research in the military is the lack of privileged communication. As a result, it is difficult to obtain valid self-reports due to a tendency to deny or minimize use. The investigators recently developed and validated a method for collecting anonymous data over time. This will be the first study in the military, as well as the first large scale, adequately powered trial, where intervention effects will be tracked out to a 6-month follow-up. The study's Specific Aims are to randomize approximately 3000 Airmen to either the current BAI versus the BAI+Text messages timed to occur before, during, and after Airmen have access to alcohol; and to evaluate the efficacy of the intervention at the end of training and 6 months post-training using repeated surveys with unique identifiers allowing researchers to match surveys while maintaining anonymity.

DETAILED DESCRIPTION:
Episodic heavy or binge drinking and the associated health and social consequences are substantial public health concerns, with a high prevalence among young adults. This is particularly true among US military personnel. While alcohol consumption in the US military is very high and normative, there is zero tolerance for getting in legal trouble while drinking, and Airmen who do get in alcohol-related legal trouble (e.g., DUI, sexual assault) typically receive what is called an Alcohol Related Incident (ARI).

In other populations, Brief Alcohol Interventions (BAIs) for alcohol misuse have been validated as efficacious with robust evidence for mostly college young adults who report episodic heavy drinking. Many BAI studies have targeted young adults who drink hazardously; these individuals are generally not interested in abstaining from alcohol but are often willing to decrease the amount they drink or change the manner in which they drink in order to reduce harmful consequences. The investigators have previously published the results of a BAI group-based intervention that has been shown to reduce ARIs universally (not in just high-risk drinkers) in over 150,000 on average by 16%. Since this intervention began in 2010, the BAI has been disseminated to most Airmen in Technical (Advanced) Training in the US Air Force. However, it is clear that additional research is needed to enhance the efficacy of the BAI intervention and to reduce the risk associated with problem drinking behavior. One such strategy that could improve health promotion outcomes is well timed and tailored automated text messages. Building on the preliminary study where text messages reduced driving after drinking as well as total drinks consumed before driving, text messaging may be highly effective as the precise time that Airmen gain access to alcohol (when they are allowed off base for the first time) is known and is the same time point for all Airmen.

One of the challenges to conducting alcohol research in the military is the lack of privileged communication. As a result, it is difficult to obtain valid self-reports due to a tendency to deny or minimize use. Fortunately, the research team has recently validated a method for collecting anonymous data over time.

This study will randomize approximately 3000 Airmen to either the currently administered group BAI versus the BAI + Interactive Counselor Facilitated Text messages timed to occur before, during, and after Airmen have access to alcohol; and (2) To evaluate the efficacy of the intervention at an end of training and 6-month follow-up using repeated anonymous surveys with unique identifiers allowing investigators to match up surveys while simultaneously maintaining anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Must be a United States Air Force Technical Training student in one of the following training groups or wings: 37th Training Wing, 81st Training Wing, 82nd Training Wing, or 59th Training Group.
* Must be 18 years of Age
* Must be able to understand English
* Must be able to receive text messages

Exclusion Criteria:

* Under 18 years of age
* Not in the specified Technical Training groups or wings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AUDIT | Baseline, 60 days, 6 months
  The study will use the AUDIT as a measure of hazardous drinking anonymously at baseline, and at follow-ups at 60 days and 6 months post intervention.
Daily Drinking Questionnaire with NIAAA recommended assessment items | Baseline, 60 days, 6 months
  The study will use this tool to measure the number of drinks per week anonymously at baseline and at follow-ups at 60 days and 6 months. This includes the NIAAA recommended alcohol assessment items. A binge episode will be SAMHSA's definition as 5 or more alcoholic drinks for males or 4 or more alcoholic drinks for females within a 2-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Kara P Wiseman, MPH, PhD, Principal Investigator — University of Virginia
Locations (1):
- JBSA Lackland, San Antonio, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT06318975/ICF_000.pdf